CLINICAL TRIAL: NCT01356225
Title: A Randomized, Double-blind, Placebo-controlled, Parallel, Single-dose Study of Intranasal Ketorolac in the Treatment of Pain Secondary to Dental Impaction Surgery
Brief Title: A Single-dose Study of Intranasal Ketorolac in the Treatment of Pain Secondary to Dental Impaction Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: David Bregman, M.D., Ph.D., Luitpold Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROX 2003-05
Record Dates: First submitted 2011-05-16; First posted 2011-05-19 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Pain; Dental Impaction
Keywords: pain following dental impaction surgery
MeSH Terms: conditions — Pain; Tooth, Impacted | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intranasal Ketorolac tromethamine (Experimental)
  Interventions: Drug: Ketorolac tromethamine
- Intranasal placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac tromethamine — 30 mg Intranasal (2 x 100 uL of a 15% solution), single dose
  Arms: Intranasal Ketorolac tromethamine
Drug: Placebo — IN placebo
  Arms: Intranasal placebo

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy of a single intranasal (IN) administration of ketorolac after dental impaction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 18 years or older.
* Body weight > or = to 100 pounds and < or = 300 pounds.
* Women of childbearing potential must have a negative serum pregnancy test result prior to entry into the study.
* Able to provide written informed consent.
* At least moderate pain as determined by a PI score of > or = to 50 mm on a 100-mm VAS.
* Willing and able to comply with all testing and requirements defined in the protocol.
* Willing and able to complete the posttreatment visit.
* Immediately prior to entering the study, surgical removal of 3 or 4 third molars (at least 1 mandibular partial bony or complete bony impaction).

Exclusion Criteria:

* Allergy or sensitivity to ketorolac or EDTA.
* Allergic reaction to aspirin or other NSAIDs.
* Current upper respiratory tract infection or other respiratory tract condition that could interfere with the absorption of the nasal spray or with the assessment of adverse events (AEs).
* Use of any IN product within 24 hours prior to study entry.
* Clinically significant abnormality on screening laboratory tests.
* History of cocaine use resulting in nasal mucosal damage.
* Active peptic ulcer disease, recent (defined as within 6 months) history of peptic ulcer disease or gastrointestinal bleeding considered by the investigator to be clinically significant.
* Advanced renal impairment (serum creatinine >1.5 mg/dL) or a risk for renal failure due to volume depletion.
* A history of any other clinically significant medical problem, which in the opinion of the investigator would interfere with study participation.
* Participation within 30 days of study entry or within 5 times the half- life, whichever is longer, in another investigational drug study.
* Pregnancy or breastfeeding.
* Extraction of teeth other than third molars during the surgical procedure; exceptions:(1) supernumerary third molars; (2) cases whereby extraction of a third molar requires the removal of an adjacent molar.
* Previous participation in this study.
* Use of any short-acting NSAID (such as aspirin or ibuprofen) or acetaminophen within 12 hours of surgery.
* Use of longer-acting NSAIDs (such as naproxen sodium) within 48 hours of surgery or piroxicam within 7 days of surgery.
* Use of steroids (other than oral contraceptives) within 72 hours of surgery.
* Use of mood-altering drugs, such a cannabis or alcohol, within 12 hours of surgery.
* Surgical anesthesia including narcotic agents except fentanyl. Short-acting anesthetics, both DEA scheduled and unscheduled, were allowed. Naloxone in any form was not permitted.
* Use of any other medication within 24 hours prior to surgery that, in the opinion of the investigator, could confound the subject's efficacy assessments (eg, sedatives, tranquilizers, MAO inhibitors, phenothiazines).
* Consumption of any caffeine-containing products within 4 hours of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-02; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference (SPID) | 8 hours postdose
  Ratings of Pain Intensity (PI) were made using a 100-mm Visual Analog Scale (VAS) on which 0 = no pain and 100 = worst pain possible. The PI values were obtained at 20 and 40 minutes, and at 1, 1.5, 2, 3, 4, 5, 6, 7, and 8 hours following the first dose of study medication on Day 1. Pain intensity difference (PID) was calculated by subtracting the posttreatment score from the baseline score, where the baseline score was the PI rating made prior to the first dose of study medication. A summed PID (SPID) on the first postoperative day was calculated at 8 hours.

SECONDARY OUTCOMES:
Summed Pain Intensity Difference (SPID) | 4 and 6 hours postdose
  Ratings of Pain Intensity (PI) were made using a 100-mm Visual Analog Scale (VAS) on which 0 = no pain and 100 = worst pain possible. The PI values were obtained at 20 and 40 minutes, and at 1, 1.5, 2, 3, 4, 5, 6, 7, and 8 hours following the first dose of study medication on Day 1. Pain intensity difference (PID) was calculated by subtracting the posttreatment score from the baseline score, where the baseline score was the PI rating made prior to the first dose of study medication. A summed PID (SPID) on the first postoperative day was calculated at 4 and 6 hours.
Total Pain Relief (TOTPAR) | 4, 6, and 8 hours postdose
  Scores were obtained from the pain relief evaluations by taking a weighted sum of pain relief scores. Pain relief was measured at 20 and 40 minutes, and at 1, 1.5, 2, 3, 4, 5, 6, 7, and 8 hours on a 5-point categorical scale where 0 = no pain relief, 1 = a little pain relief, 2 = some pain relief, 3 = a lot of pain relief, and 4 = complete pain relief.
Pain intensity difference (PID) and pain relief scores | Before receiving study drug (baseline), at 20 and 40 minutes, and at 1, 1.5, 2, 3, 4, 5, 6, 7, and 8 hours postdose
  Ratings of Pain Intensity (PI) were made using a 100-mm Visual Analog Scale (VAS) on which 0 = no pain and 100 = worst pain possible. PID was calculated by subtracting the posttreatment score from the baseline score, where the baseline score was the PI rating made prior to the first dose of study medication. Pain relief was measured on a 5-point categorical scale with 0 = no pain relief, 1 = a little pain relief, 2 = some pain relief, 3 = a lot of pain relief, and 4 = complete pain relief.
Peak PID score | 4, 6, and 8 hours postdose
  PID was calculated by subtracting the posttreatment score from the baseline score, where the baseline score was the PI rating made prior to the first dose of study medication. Peak PID was defined as the maximum PID score.
Peak pain relief scores | 4, 6, and 8 hours postdose
  Pain relief was measured on a 5-point categorical scale with 0 = no pain relief, 1 = a little pain relief, 2 = some pain relief, 3 = a lot of pain relief, and 4 = complete pain relief. Peak pain relief was defined as the maximum peak pain relief score.
Time to onset of perceptible pain and meaningful pain relief | After study drug administration until perceptible and meaningful pain relief was felt (during the 8-hour postdose observation period)
  The onset of pain relief was measured by the subjects stopping stopwatches when perceptible and meaningful relief was felt.
Time to first use of rescue medication | After study drug administration until rescue analgesic therapy was requested (during the 8-hour postdose observation period)
  Duration of analgesia represented by the time until rescue analgesic therapy was requested.
Proportion of subjects taking rescue medication | During 8-hour postdose observation period
  Proportion of subjects taking rescue medication in either group during the 8-hour postdose observation period.
Global pain control | At the end of the 8-hour observation period, or at the time the subject took rescue analgesic medication if prior to 8 hours
  The subject was asked the question "How was your pain control overall?" This evaluation was measured on a 5-point categorical scale with 0 = poor, 1 = fair, 2 = good, 3 = very good, and 4 = excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Lincoln Bynum, MD, Study Chair — GloboMax (ICON plc)
Locations (1):
- Austin Oral Surgery - PPD Development, Austin, Texas, United States